CLINICAL TRIAL: NCT01798264
Title: A Phase Ib, Randomized, Open-Label, Multi-Center, 4-Week Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ITCA 650 in Subjects With Type 2 Diabetes Mellitus
Brief Title: Open Label, 4 Week Study of ITCA 650 in Adults With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITCA 650-CLP-01
Record Dates: First submitted 2013-02-20; First posted 2013-02-25 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

ARMS (4):
- 10 mcg./day (Experimental): ITCA 650 (exenatide in DUROS)
  Interventions: Drug: ITCA 650 (exenatide in DUROS)
- 20 mcg/day (Experimental): ITCA 650 (exenatide in DUROS)
  Interventions: Drug: ITCA 650 (exenatide in DUROS)
- 40 mcg/day (Experimental): ITCA 650 (exenatide in DUROS)
  Interventions: Drug: ITCA 650 (exenatide in DUROS)
- 80 mcg/day (Experimental): ITCA 650 (exenatide in DUROS)
  Interventions: Drug: ITCA 650 (exenatide in DUROS)

INTERVENTIONS:
Drug: ITCA 650 (exenatide in DUROS)

SUMMARY:
evaluate the safety and tolerability of ITCA 650 in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes >6 months
* stable diet & exercise, metformin, TZD or met + TZD HbA1c >6.5% <10.0%

Exclusion Criteria:

* prior treatment with exenatide
* history of pancreatitis
* history of medullary thyroid cancer or multiple endocrine neoplasia 2

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Miami Gardens, Florida
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio
  - dGd Research, San Antonio, Texas

REFERENCES:
- [Derived] Henry RR, Logan D, Alessi T, Baron MA. A randomized, open-label, multicenter, 4-week study to evaluate the tolerability and pharmacokinetics of ITCA 650 in patients with type 2 diabetes. Clin Ther. 2013 May;35(5):634-645.e1. doi: 10.1016/j.clinthera.2013.03.011. Epub 2013 Apr 8. PMID 23578605

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initiated February 2009 completed 15 May 2009
Groups:
- 10 Mcg/Day; 20 Mcg/Day; 40 Mcg/Day; 80 Mcg/Day: ITCA 650 (exenatide in DUROS)
Period: Overall Study
Arm/Group | 10 Mcg/Day | 20 Mcg/Day | 40 Mcg/Day | 80 Mcg/Day
Started | 12 | 11 | 10 | 11
Completed | 11 | 11 | 10 | 7
Not Completed | 1 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 Mcg/Day | 20 Mcg/Day | 40 Mcg/Day | 80 Mcg/Day | Total
Number analyzed (Participants) | 12 | 11 | 10 | 11 | 44
Age Continuous [Mean (Standard Deviation); unit: years] | 56.3 (6.74) | 57.2 (6.10) | 52.6 (9.54) | 56.5 (4.84) | 55.7 (6.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 6 | 4 | 18
  Male | 8 | 7 | 4 | 7 | 26
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 10 | 11 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Study Drug-Related Adverse Events
Time Frame: 4 weeks
Population: Number of subjects reporting study drug-related adverse events
Measure: Number; unit: participants
Arm/Group | 10 Mcg/Day | 20 Mcg/Day | 40 Mcg/Day | 80 Mcg/Day
Number analyzed (Participants) | 12 | 11 | 10 | 11
participants | 9 | 11 | 9 | 11

2. Secondary Outcome: To Characterize the Pharmacokinetic Profile of ITCA 650 in Subjects With Type 2 Diabetes Mellitus
Description: Change in HbA1c from baseline
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 10 Mcg/Day | 20 Mcg/Day | 40 Mcg/Day | 80 Mcg/Day
Number analyzed (Participants) | 12 | 11 | 10 | 11
percentage | -0.5 (0.39) | -0.6 (0.31) | -0.5 (0.31) | -0.7 (0.36)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) 4 Weeks From Baseline
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 Mcg/Day | 20 Mcg/Day | 40 Mcg/Day | 80 Mcg/Day
Number analyzed (Participants) | 12 | 11 | 10 | 11
mg/dL | -5.6 (34.33) | -31.2 (24.2) | -42.0 (33.16) | -28.8 (33.5)

4. Secondary Outcome: Change in Weight From Baseline to 4 Weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 10 Mcg/Day | 20 Mcg/Day | 40 Mcg/Day | 80 Mcg/Day
Number analyzed (Participants) | 12 | 11 | 10 | 11
kg | -0.3 (0.91) | -0.3 (1.51) | -1.1 (1.6) | -3.1 (2.13)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | 10 Mcg/Day | 20 Mcg/Day | 40 Mcg/Day | 80 Mcg/Day
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 12/12 | 11/11 | 9/10 | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 Mcg/Day (N=12) | 20 Mcg/Day (N=11) | 40 Mcg/Day (N=10) | 80 Mcg/Day (N=11)
eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 6 (9) | 8 (23)
vomiting (Gastrointestinal disorders) | 0 (0) | 3 (6) | 1 (5) | 9 (23)
dyspepsia (General disorders) | 0 (0) | 1 (1) | 1 (2) | 4 (5)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
abdominal disomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
GERD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
early satiety (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
incision site erythema (Injury, poisoning and procedural complications) | 4 (6) | 6 (9) | 6 (16) | 5 (11)
incision site complication (Injury, poisoning and procedural complications) | 6 (8) | 7 (8) | 7 (16) | 5 (8)
incision site hemmorhage (Injury, poisoning and procedural complications) | 3 (4) | 5 (6) | 2 (4) | 3 (4)
incision site pain (Injury, poisoning and procedural complications) | 4 (5) | 1 (3) | 2 (3) | 5 (6)
incision site blister (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 4 (6) | 2 (2)
incision site edema (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 3 (3) | 6 (6)
hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
hyperamylasemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 1 (2) | 1 (1) | 2 (2) | 2 (5)
dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (3)
paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
dizziness extertional (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days